CLINICAL TRIAL: NCT02097082
Title: An Evaluation of the 480 Biomedical STANZA™ Drug-Eluting Resorbable Scaffold (DRS) System in the Treatment of de Novo SFA Lesions
Brief Title: Treatment of SFA Lesions With 480 Biomedical STANZA™ Drug-Eluting Resorbable Scaffold (DRS) System
Acronym: SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 480 Biomedical (Industry)
Responsible Party: Sponsor
Organization: Lyra Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 480-SFA2013-001
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases
Keywords: Peripheral Arterial Disease; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases; Superficial Femoral Artery
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STANZA Drug-eluting Resorbable Scaffold (Experimental): Treatment of Superficial Femoral Artery (SFA) lesion with resorbable scaffold
  Interventions: Device: STANZA Drug-eluting resorbable Scaffold

INTERVENTIONS:
Device: STANZA Drug-eluting resorbable Scaffold
  Other Names: Paclitaxel-eluting resorbable scaffold

SUMMARY:
An evaluation of the safety and performance of the STANZA Drug-eluting Resorbable Scaffold (DRS) system for the treatment of patients with obstructive superficial femoral artery disease.

DETAILED DESCRIPTION:
The STANZA DRS system is comprised of a controlled release paclitaxel-eluting bioresorbable scaffold and a delivery system used in the treatment of superficial femoral artery disease.

ELIGIBILITY:
Inclusion Criteria

1. Age > 18 years.
2. De novo stenotic lesion(s) in the superficial femoral artery located at least 1 cm distal to the femoral bifurcation and > 5 cm above the joint space of the knee.
3. Patient has symptomatic intermittent claudication affecting at least the target leg (Rutherford Class 2-3). Patients should have first received conservative medical management of their symptoms prior to study inclusion. The symptoms can be bilateral.
4. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the ethics committee of the respective clinical site.
5. The study patient agrees to comply with all required post-procedure study requirements.

Baseline Inclusion Criteria

1. Reference vessel diameter (RVD) 5.0 -6.0 mm measured by an objective measurement such as online Quantitative Vessel Analysis (QVA).
2. Target lesion length ≤ 90 mm; total occlusion length < 40 mm.
3. Target lesion has a ≥70% diameter stenosis.
4. Angiographic evidence of at least one runoff vessel to the ankle/foot without hemodynamically significant stenosis (>50% diameter stenosis) that does not require any treatment within 3 months of the index procedure.
5. Procedural access can be accomplished via contralateral vascular access or if antegrade access no closure device can be utilized and closure has to occur via manual pressure.
6. Patent common and external iliac: TASC A & B iliac lesions may be treated at the time of index procedure (before treatment of the target lesion) if residual stenosis is ≤30%.

Exclusion Criteria

1. Previous vascular surgery/endovascular treatment of the target lesion.
2. Re-vascularization of target vessel within 30 days of study procedure.
3. Critical limb ischemia defined as Rutherford Becker Category 4-6.
4. Known coagulation disorders or intolerance or allergies to aspirin, clopidogrel or ticlopidine, heparin, any scaffold components, contrast agents which cannot be adequately pre-medicated.
5. Life expectancy ≤12 months.
6. Planned procedure that necessitates the discontinuation of antiplatelet medications used in conjunction with the investigational device within 3 months post-procedure.
7. Inability to walk due to orthopedic or other nonvascular complications.
8. Pregnancy or breast feeding or patient desires to become pregnant.
9. Non-atherosclerotic lesion (e.g. vasculitis).
10. Renal insufficiency (serum creatinine level > 220 µmol/L or > 2.5 mg/dl, or patient is on dialysis).
11. Patient has medical condition(s) which could affect study assessments or may adversely affect the safety and/or success of the study treatment.
12. Active systemic infection or lower limb infection of any nature.
13. White Blood Cells (WBC) ≤ 3,000 cells/mm3.
14. Myocardial infarction within 30 days prior to the study procedure.
15. Stroke within 90 days prior to the study procedure.
16. Uncontrolled atrial fibrillation.
17. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
18. Prior use of paclitaxel-eluting products in the target limb less than 6 months prior to index procedure.
19. Patient has known unstable angina.

Baseline Exclusion Criteria

1. Target lesion treatment with a drug eluting balloon.
2. Target lesion treatment with atherectomy, laser, or cryoplasty (use of a cutting or scoring balloon is permitted prior to scaffold implantation only).
3. Suspicion for or evidence of subintimal passage of guidewire.
4. Severely calcified lesion(s).
5. Target lesion which, based on two angiographic orthogonal views, exhibit a persistent balloon deformity during pre-dilatation with a nominally sized balloon.
6. Target vessel (superficial femoral artery) has an angiographically significant (> 50% diameter stenosis) lesion located distally or proximally to the target lesion.
7. Acute embolic complication following pre-dilatation.
8. Target vessel contains an acute thrombus.
9. Aneurysm in target vessel or co-existing clinically significant aneurysmal disease of the abdominal aorta, iliac or popliteal arteries.
10. Intervention in the infra-inguinal arteries outside of the target lesion.
11. Planned procedure within 30 days after the index procedure.
12. Positive pregnancy test for females of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03-30 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Patency by Ultrasound | through 6 months
  Patency measured by duplex ultrasound with ≤50% restenosis (Peak Systolic Velocity Ratio (PSVR ≤ 2.4).
Major Adverse Events | 30 days
  Freedom from all causes of death, emergent endovascular intervention or surgical intervention on the target limb, index limb amputation.

SECONDARY OUTCOMES:
Clinical Success | 48 hours
  On a per patient basis, technical success without major adverse event (MAE) within 48 hours after the index procedure or at hospital discharge, whichever is sooner.
Device Success | Procedure
  On a per device basis, the achievement of successful delivery and deployment of the study device at the intended target lesion and successful withdrawal of the delivery catheter.
Technical Success | Procedure
  Technical success is defined on a per lesion basis, as the achievement of a final residual stenosis of ≤ 30%.
Patency by Ultrasound | 12, 24 months
  Patency measured by duplex ultrasound with ≤50% restenosis (PSVR ≤ 2.4) based on core lab evaluation at 12 and 24 months.
Patency by Angiography | 12 months
  ≤50% diameter stenosis determined by an angiographic core lab analysis of an angiogram performed at 12 months.
Clinically Driven Target Lesion Revascularization (TLR) | 6,12, 24 months
  Clinically Driven TLR is defined as symptomatic patients with:
  Decrease in Ankle Brachial Index (ABI) > 0.15 and Increase in Rutherford Becker Category ≥ 1 from post procedure assessment and >50% stenosis by angiography.
Surgical Intervention on the target limb, index limb amputation | 3,6,12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (9):
- Austria (3):
  - Universitäts Klinikum Graz, Graz
  - WGKK - Hanusch-Krankenhaus, Vienna
  - Cardiovascular and Interventional Radiology- AKH, Vienna
- Germany (3):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen GmbH, Bad Krozingen, Baden-Wurttemberg
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
- Auckland City Hospital, Auckland, New Zealand
- Switzerland (2):
  - INSELSPITAL, Universitätsspital Bern, Bern
  - University Hospital Zurich, Zurich